CLINICAL TRIAL: NCT06688149
Title: NASH Patient's Itinerary: Comparison of Strategies for Screening, Referring and Management of Diabetic Patients
Acronym: NASH-PI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Collaborators: Gilead Sciences (Industry); Barcelona Institute for Global Health (Other); Harokopio University (Other); University Medical Center Mainz (Other); University Düsseldorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: NASH-PI
Record Dates: First submitted 2024-10-30; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD)
Keywords: NAFLD; MASLD; NASH; MASH; FIBROSIS; NITs; TRANSIENT ELASTOGRAPHY; FIB4; NFS; HFS; DIABETES
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: Current management of NAFLD patients in daily clinical practice (Experimental): It will be taken as a reference for comparisons and will include the diagnosis and referral criteria that have been used the two previous years. CONSTANTS, a study included in the EPOS European Project has already allowed us to approach the burden of this entity in clinical practice in two sites of this consortium (Mainz and Sevilla). An overall analysis will be conducted to harmonize current standard of care (Arm A) in our centres. The case records of all patients referred with a diagnosis of NAFLD will be reviewed and evaluated for evidence of advanced fibrosis/cirrhosis based on a composite of history, physical examination, imaging, transient elastography, and liver histology when available. HFS, NFS, and FIB-4 scores will be calculated, and patients with a priori low-risk of advanced fibrosis will be deemed to have no evidence of liver fibrosis and thus referred inappropriately.
  Interventions: Diagnostic Test: Derivation algorithms
- Arm B: Combination of blood-based non-invasive tests (HFS, NFS, and FIB-4) (Experimental): Patients will be assigned with the following scores:
  1. 0 points if the value is under the lower cut-off (HFS <0.12; NFS<-1.455; FIB-4 <1.30);
  2. 1 point if the value is allocated in the grey zone (HFS 0.12-0.47; NFS -1.455-0.676; FIB-4 1.30-2.67);
  3. 2 points if the value is above the higher cut-off (HFS >0.47; NFS >0.676; FIB-4 >2.67). We will determine the optimal cut-offs (between 0 and 6 points) for keeping patients in non-specialized units or referring them to NSUs.
     * Age corrected threshold should be implemented in patients older than 65 years in NFS (from -1.455 to 0.12) and FIB-4 (from 1.30 to 2.00).
  Interventions: Diagnostic Test: Derivation algorithms
- Arm C: Combination of HFS and TE (Experimental): Patients will be classified using the blood-based non-invasive tests to determine the HFS and a transient Elastography (TE). Patients with a HFS score of > 0.12 or TE >8 kPa for both M and XL probe should be classified as patients with an intermediate-to-high risk of advanced fibrosis and will be referred to a specialist.
  Interventions: Diagnostic Test: Derivation algorithms

INTERVENTIONS:
Diagnostic Test: Derivation algorithms — Derivation algorithm based on non-invasive methods, to standardise the continuum of care for diabetic patients with NAFLD from primary care and endocrinology settings to NAFLD specialised units (NSU)

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is a highly prevalent, underdiagnosed, health system burden and impacts on quality of life including comorbidities in the affected population. Cost-effective strategies focusing on clinical pathways to detect and refer patients to care are needed. The aim of this study is to build a stepwise algorithm combining non-invasive freely available methods (FIB-4, NFS, HFS alone or combined) and vibration-controlled transient elastography (VCTE) in diabetic patients from primary care and endocrinology units.

DETAILED DESCRIPTION:
NAFLD is a growing health concern and liver fibrosis severity determines its prognosis. The burden of this disease has been estimated in a quarter of the European population and is even higher in diabetic patients, where it raises significantly and can reach up to 80%. The fact that only 10% of these patients will develop significant fibrosis, the strongest predictor of liver-specific morbidity and overall mortality, leads to an overwhelming situation in primary care and endocrine units, where physicians need to screen large numbers of patients to identify individuals with a high risk for developing fibrosis that should be derived to a specialized hepatology unit. New free and accurate non- invasive tests need to be available to be used in primary care and non-hepatologists units to fight against this disappointing situation.

Several non-invasive methods, based on serum and imaging biomarkers, have aimed to identify at-risk patients for NAFLD-related fibrosis, but inconclusive results and many phenotypes that are present or not in patients (diabetes mellitus, obesity and age) reduce their diagnostic accuracy. Current strategies to monitor fibrosis are, therefore, inefficient and often fail to easily distinguish patients with mild disease that can be monitored at primary care from those at risk of advanced fibrosis or cirrhosis that need to receive specialised care and that could benefit from therapeutic interventions, such as participation in clinical trials and liver cancer surveillance programs.

The majority of patients with NAFLD are followed up in the community by general practitioners without definite diagnosis, representing a challenge to identify patients at risk of significant fibrosis who might benefit from an early specific intervention. Accurate fibrosis assessment by primary care or non-hepatologists physicians is limited by a reliance on liver function tests, which correlate poorly with fibrosis, and limited access to discriminatory fibrosis tests. Thus, current management strategies are inefficient in identifying subjects for specialist referral. Patients with mild disease are often referred for NAFLD specialist review when instead the appropriate preventative interventions of lifestyle changes can be delivered effectively in primary care. Conversely, patients with advanced fibrosis or cirrhosis who will benefit from NAFLD specific interventions, including clinical trials and cirrhosis surveillance, often remain undetected until they present with complications of cirrhosis, including hepatocellular carcinoma. This ineffective management contributes to the poor outcomes associated with liver disease and the increasing trends in NAFLD- related morbidity and mortality.

NASH-PI aims to improve the management of NAFLD patients by non-hepatologist physicians through the development of a new specific stepwise NAFLD algorithm following an ETC (Education, tools and communication) process that will be based on:

1. The development of new care pathways based on different combinations of non-invasive tests that facilitate the derivation of diabetic patients from endocrine and primary care units to specialised liver disease units.
2. Peer-to-peer sessions with primary care physicians and diabetologists to discuss the techniques and methods available to screen and detect diabetic patients at risk of developing NAFLD-related significant fibrosis.
3. The implementation of easy and ready to use tools, like an automatic calculation of fNITs in central labs, to allow non-hepatologist physicians detect more efficiently diabetic patients at risk of significant fibrosis.

This proposal will focus on diabetic patients to test the feasibility and accuracy of these diagnostic strategies in a close circuit from primary care and diabetic clinics to NAFLD specialized Units (NSU). Our main goal is to create a NAFLD continuum of care that improves the selection of patients with fibrosis and cirrhosis for referral to secondary care, reducing unnecessary referrals, enhancing the use of healthcare resources with immediate cost-savings, and improving patient experiences by avoiding unnecessary clinic appointments and tests. NASH-PI will improve the identification of NAFLD in diabetic patients to allow for management according to current standard of care and impact on the disease course, helping to reduce NAFLD-related morbidity and mortality and delivering more efficient patient-centered care.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75.
2. Type 2 Diabetes Mellitus. Patients will be considered as diabetic when: A1C ≥6.5% OR FPG ≥126 mg/dL OR 2-h PG ≥200 mg/dl during the OGTT OR anti-diabetic drug users.

Exclusion Criteria:

1. Significant alcohol intake (>30 g daily for men and >20g daily for women).
2. Evidence of concomitant liver disease (i.e., viral or autoimmune hepatitis, HIV, drug-induced fatty liver, hemochromatosis, or Wilson's disease).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 536 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2024-01-08 (Actual)

PRIMARY OUTCOMES:
Accuracy on referral rate | Up to 6 months
  To determine the accuracy on referral rate for diabetic patients at risk of advanced fibrosis using each of the strategies under study, and determine the sensitivity, specificity, PPV, NPV, likelihood ratios and overall accuracy of each of them.

SECONDARY OUTCOMES:
Cut-off scores for fibrosis non-invasive tests (fNITs) | 3 months
  To define the best cut-off scores for fibrosis non-invasive tests (fNITs) when all these non-invasive tests are combined between them. Combined fibrosis score is a composite score including the results from FIF4, HFS and NFS, and ranges from 0 (no risk of fibrosis) and 3 (all 3 tests are altered and therefore patients have from more than 90% of risk of fibrosis).
Cut-off score for Hepamet Fibrosis Score (HFS) + Transient Elastography (TE) | 3 months
  To define the best cut-off score for the Hepamet Fibrosis Score (HFS) when combined with Transient Elastography (TE). HFS higher that 0.12 indicates high risk of liver fibrosis, and TE higher that 8 KPa indicates risk of significant liver fibrosis.
Evaluation of quality-adjusted life years (QALYs) | 9 months
  QALY scores will compare the benefits of the 3 different strategies/arms. QALY = Life Years Gained × Quality of Life Score. Quality of Life Score will be calculated by the Short-Form Six-Dimension (SF-6D) questionnaire, and ranges from 1 (perfect health) to 0 (death).
Evaluation of Incremental Cost-Effectiveness Ratios (ICERs) | 9 months
  ICER will assess the cost per additional unit of health benefit achieved with each of the 3 strategies under study, calculated as euros per QALYs gained.
Patient reported diet habits | 6 months
  To assess patient reported diet habits by the PREDIMED questionnaire, a validated 14-item questionnaire of Mediterranean diet adherence. Score lower than 9 means low adherence to Mediterranean diet, and score equal or higher than 9 means good adherence to Mediterranean diet
Patient reported physical activity | 6 months
  To assess patient reported physical activity using the International Physical Activity Questionnaire (IPAQ) questionnaire. IPAQ classifies individuals into three categories based on their total Metabolic Equivalent of Task (MET) minutes per week. Low physical activity: Less than 600 MET-minutes/week; moderate physical activity: Between 600 and 3,000 MET-minutes/week; or high physical activity: More than 3,000 MET-minutes/week.
Patient reported individual functioning | 6 months
  To assess patient reported individual functioning by the Short-Form Six-Dimension (SF-6D) questionnaire. Scores Closer to 1 indicate better health-related quality of life. Scores Closer to 0 reflect more severe health problems and limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Romero-Gómez, Principal Investigator — Hospital Universitario Virgen del Rocío de Sevilla
Locations (4):
- Germany (2):
  - University Hospital Düsseldorf, Düsseldorf
  - University Medical Center Mainz, Mainz
- Harokopio University of Athens, Athens, Greece
- Hospital Universitario Virgen del Rocío de Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: No